CLINICAL TRIAL: NCT02417103
Title: Pretreatment of Patients Expecting Bariatric Surgery With the GLP-1 Analogon
Brief Title: Pretreatment of Patients Expecting Bariatric Surgery With the GLP-1 Analogon Liraglutid
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruiting failure
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLP1Bariatric
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucagon-Like Peptide 1; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLP-1 (Liraglutide) (Active Comparator): Daily subcutaneous injection of Lirglutide over 9 weeks prior to bariatric surgery with a dosing of 0,6-1,8 mg
  Interventions: Drug: GLP-1 (Liraglutide)
- Placebo Comparator (Placebo Comparator): Daily subcutaneous injection of PL1/PR1 Placebo over 9 weeks prior to bariatric surgery with a dosing of 0,6-1,8 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLP-1 (Liraglutide) — GLP-1 Analogon
  Other Names: Victoza
  Arms: GLP-1 (Liraglutide)
Drug: Placebo — Placebo
  Other Names: PL1 PR1
  Arms: Placebo Comparator

SUMMARY:
The aim of this study is to investigate the effect of the treatment with the GLP-1 Analogon Liraglutide on the lipid metabolism an inflammation in adipose tissue.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of the treatment with the GLP-1 Analogon Liraglutide on the lipid metabolism an inflammation in adipose tissue. As GLP-1 is presumed to improve insulin sensitivity and associated parameters the investigators hypothesize that this might be due to changes in lipid metabolism which might be involved in the regulation of insulin sensitivity. Therefore the investigators intend to investigate changes of metabolic pathways before and after treatment with the GLP-1 analog liraglutide that could play a crucial role in pathogenesis as well as regulation of insulin sensitivity and atherogenic dyslipidemia such as: de novo lipogenesis and reverse cholesterol transport

ELIGIBILITY:
Inclusion Criteria:

* BMI 35-55 Kg/m2
* Fasting Blood glucose >140mg/dl
* Planned bariatric surgery
* Diabetic Medication (Metformin, Sulfonylurea, Insuline)

Exclusion Criteria:

* Known hypersensitivity against Liraglutid
* Pretreatment DPP-4 Inhibitors or GLP-1 Analogue the last 3 months
* HbA1c >10%

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
weight reduction | 4 years
  to compare body weight with type 2 Diabetes scheduled for weight loss surgery after 8 weeks of preoperative treatment with either placebo or liragludite

SECONDARY OUTCOMES:
GLP-1 Levels | 4 years
  Measurement of GLP-1 levels during the defined period

CONTACTS AND LOCATIONS:
Overall Officials: Jens Aberle, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg, Hamburg, Germany